CLINICAL TRIAL: NCT03707171
Title: Effects of Liraglutide on the Cognitive Function in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of the department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Liraglutide
Record Dates: First submitted 2018-09-27; First posted 2018-10-16 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Cognitive function; Liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide (Active Comparator): 12 weeks of liraglutide treatment at adjusting dose, up to 1.8mg/day Drug: liraglutide
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): 12 weeks of Placebo treatment at adjusting dose Drug:Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Liraglutide — Liraglutide is a glucagon-like peptide type 1 (GLP-1) analogue. It has been proved that Liraglutide can improve insulin resistance and cognitive function in AD animals. Therefore, it is speculated that Liraglutide may interfere with the occurrence and development of cognitive dysfunction in patients with T2DM. In order to confirm the effects, the investigators conduct an open, prospective, positive controlled study in patients with T2DM.
  Arms: Liraglutide
Drug: placebo — Any hypoglycemic drugs except glucagon-like peptide type 1 (GLP-1) analogue.
  Arms: Placebo

SUMMARY:
Type 2 diabetes mellitus (T2DM) can impaire cognitive function,the prevalence of Alzheimer's Disease(AD) in T2DM patients is 1.5 to 2.5 times higher than the general population.Cognitive impairment seriously affects the health and quality of life of the elderly. Prevention and treatment measures for cognitive decline in persons with T2DM has not been well studied.

Glucagon-like peptide-1 (GLP-1) is a member of an endogenous class of incretin hormones synthesized in intestinal epithelial L-cells.GLP-1 enhances glucose-dependent secretion of insulin,inhibits glucagon secretion, slows gastric emptying and reduces food intake. Liraglutide is a glucagon-like peptide type 1 (GLP-1) analogue. It has been proved that Liraglutide can improve insulin resistance and cognitive function in AD animals. Therefore, it is speculated that Liraglutide may interfere with the occurrence and development of cognitive dysfunction in patients with T2DM. In order to confirm the effects, the investigators conduct an open, prospective, positive controlled study in patients with T2DM. The effect on BMI,waist circumference, hip circumference, waist-to-hip ratio,fasting plasma glucose，glycosylated hemoglobin,blood lipids and cognitive function were measured to explore the effects of liraglutide in patients with T2DM.

The overall goal of this study is to explore the effects of liraglutide on the cognitive function in patients with type 2 diabetes mellitus and make further contribution to the improvement of cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes。

Exclusion Criteria:

* Type 2 diabetes with acute diabetic complications.
* Type 1 diabetes.
* Other diseases affecting cognitive function (congenital dementia,brain trauma,severe heart dysfunction,severe kidney dysfunction,severe lung dysfunction,epilepsy,severe hypoglycemic coma,cerebrovascular disease,ischemic heart disease,etc).
* Alcohol abuse,mental illness and psychoactive substance abuse.
* History of thyroid disease.
* Any surgical or medical conditions that significantly influence absorption, distribution, metabolism or excretion of the intervention drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Changes of cognitive function assessed by cognitive function scale after 12 weeks. | Baseline,4weeks,8weeks，12weeks(End of Trial)
  The cognitive function will be calculated from performance on the following measures: (1)Digit Span Test(DST);(2) Rey Auditory Verbal Learning(RAVL);(3) Long-Delay Free Recall(LDFR);(4) Trail Making Test(TMT);(5) Animal Naming Test(ANT);(6) Clock Drawing Test(CDT);(7)Minimum Mental State Examination(MMSE);(8)Memory and executive screening(MES);(8)functional near-infrared spectroscopy.

SECONDARY OUTCOMES:
Changes of systolic blood pressure and diastolic blood pressure | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of systolic blood pressure and diastolic blood pressure compared with baseline, and between the intervention and control group at the end of the study (12 weeks)
Change of fasting plasma glucose | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of fasting plasma glucose compared with baseline, and between the intervention and control group at the end of the study (12 weeks)
Change of HbA1c | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of HbA1c compared with baseline, and between the intervention and control group at the end of the study (12 weeks)
Change of lipid profile | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of lipids profiles (TC, HDL-C, LDL-C, TG) in mmol/L compared with baseline, and between the intervention and control group at the end of the study (12 weeks)
Change of liver enzymes | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of liver enzymes (ALT, AST in IU/L) compared with baseline, and between the intervention and control group at the end of the study (12 weeks)
Change of kidney function | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of kidney function（serum creatinine in umol/L、eGFR in ml/min） compared with baseline, and between the intervention and control group at the end of the study (12 weeks)
Change of CRP | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of CRP compared with baseline, and between the intervention and control group at the end of the study (12 weeks)
Change of Body mass index(BMI) | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of Body mass index(BMI) compared with baseline, and between the intervention and control group at the end of the study (12 weeks)
Change of waist circumference | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of waist circumference compared with baseline, and between the intervention and control group at the end of the study (12 weeks)
Change of hip circumference | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of hip circumference compared with baseline, and between the intervention and control group at the end of the study (12 weeks)
Change of waist-to-hip ratio | Baseline,4weeks,8weeks，12weeks(End of Trial)
  Change of waist-to-hip ratio compared with baseline, and between the intervention and control group at the end of the study (12 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Li Q, Jia M, Yan Z, Li Q, Sun F, He C, Li Y, Zhou X, Zhang H, Liu X, Bu X, Gao P, He H, Zhao Z, Zhu Z. Activation of Glucagon-Like Peptide-1 Receptor Ameliorates Cognitive Decline in Type 2 Diabetes Mellitus Through a Metabolism-Independent Pathway. J Am Heart Assoc. 2021 Jul 20;10(14):e020734. doi: 10.1161/JAHA.120.020734. Epub 2021 Jul 10. PMID 34250817